CLINICAL TRIAL: NCT02089945
Title: Cognitive and Functional Outcomes Following Transcatheter Aortic Valve Implantation (TAVI): a Pilot Study
Brief Title: Pilot Study of Cognitive and Functional Outcomes Following TAVI
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 503-2013
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Aortic Stenosis
Keywords: transcatheter aortic valve implantation; severe aortic stenosis; cognition; functional capacity; quality of life
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transcatheter aortic valve implantation: This study recruits individuals that are undergoing transcatheter aortic valve implantation.

SUMMARY:
Narrowing of the aortic valve in the heart, known as severe aortic stenosis, can impede blood delivery and is associated with poor quality of life and death. In the elderly with considerable medical burden, a relatively new non-invasive valve replacement technique called Transcatheter Aortic Valve Implantation (TAVI) can be used instead of open-heart surgery. However, long term changes in cognition after TAVI remain unclear and previous studies have suggested an increased risk of cognitive decline in patients following the surgical procedure. In this pilot study, the investigators will characterize changes in cognition, physical capacity, overall quality of life and neuropsychiatric symptoms (depression and apathy) over 6 months after TAVI.

DETAILED DESCRIPTION:
Cardiovascular disease including valvular heart disease, contributes to an estimated 36% of all deaths over the age of 70. In particular, severe aortic stenosis is the most common valvular heart disease in the elderly in the Western world and is associated with reduced quality of life and increased mortality. TAVI has been shown to improve survival, with an all-cause mortality at 1 year similar to surgical aortic valve replacement (SAVR) with favourable outcomes long-term including improved functional capacity and quality of life. Recent evidence from randomized controlled trials suggests an increased risk of neurological events (e.g. cognitive decline) up to 1 year after TAVI in comparison to both SAVR and medical treatment. Studies have shown no change in short-term memory, working memory, verbal learning, delayed recognition and verbal fluency 3 months after TAVI. In addition, patients with severe aortic stenosis have an increased risk of mortality and future health complications. This study will be an observational, prospective cohort pilot study to examine changes in cognitive performance and functional outcomes after TAVI. We propose to recruit 34 patients for this study. Cognitive performance will be measured using a standardized cognitive battery prior to TAVI and 6 months post-TAVI. Functional capacity, changes in neuropsychiatric symptoms and quality of life will also be assessed prior to TAVI and 6 months post-TAVI. We hypothesize there will a change in cognitive performance, functional capacity, mood outcomes and quality of life over 6 months after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe symptomatic aortic stenosis
* undergoing TAVI
* speak and understand English

Exclusion Criteria:

* emergency TAVI
* any medical conditions that will affect their ability to complete the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of severe symptomatic aortic stenosis (aortic valve area < 1 cm2, mean gradient across the aortic valve of 40 mm Hg or more and a peak aortic jet velocity of 4.0 m/s or more) undergoing transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 6 months
  The 30-minute neuropsychiatric assessment battery recommended by NINDS-CSN (National Institute of Neurological Disorders and Stroke- Canadian Stroke Network) harmonized standards

SECONDARY OUTCOMES:
Functional capacity | 6 months
  The Timed Up and Go Test (TUG) and Hand Grip Strength Test

OTHER OUTCOMES:
Quality of life | 6 months
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) and EQ-5D-5L questionnaires
Depression | 6 months
  Centre for Epidemiologic Studies Depression Scale (CES-D)
Apathy | 6 months
  Apathy Evaluation Scale (AES)

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada